CLINICAL TRIAL: NCT02500407
Title: An Open-Label, Multicenter, Phase I/II Trial Evaluating the Safety, Efficacy, and Pharmacokinetics of Escalating Doses of Mosunetuzumab (BTCT4465A) as a Single Agent and Combined With Atezolizumab in Patients With Relapsed or Refractory B-Cell Non-Hodgkin's Lymphoma and Chronic Lymphocytic Leukemia
Brief Title: A Safety, Efficacy and Pharmacokinetic Study of BTCT4465A (Mosunetuzumab) as a Single Agent and Combined With Atezolizumab in Non-Hodgkin's Lymphoma (NHL) and Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO29781
Record Dates: First submitted 2015-07-14; First posted 2015-07-16 (Estimated); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Lymphocytic Leukemia, Chronic; Lymphoma, Non Hodgkin
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin | interventions — atezolizumab

ARMS (2):
- Dose Escalation (Experimental): Participants will receive BTCT4465A (Mosunetuzumab) via intravenous (IV) infusion or subcutaneous (SC) injection as a single-agent or in combination with atezolizumab. Dose escalation will be guided by the observed incidence of DLTs at each dose level.
  Interventions: Drug: BTCT4465A (Mosunetuzumab) IV; Drug: Atezolizumab; Drug: BTCT4465A (Mosunetuzumab) SC
- Dose Expansion (Experimental): Participants will receive BTCT4465A (Mosunetuzumab) as a single-agent or in combination with atezolizumab.
  Interventions: Drug: BTCT4465A (Mosunetuzumab) IV; Drug: Atezolizumab; Drug: BTCT4465A (Mosunetuzumab) SC

INTERVENTIONS:
Drug: BTCT4465A (Mosunetuzumab) IV — Participants with B-cell NHL and CLL will receive BTCT4465A (Mosunetuzumab) via IV infusion.
Drug: Atezolizumab — Participants assigned to an atezolizumab combination group will receive atezolizumab 1200 mg administered as an IV infusion in combination with BTCT4465A (Mosunetuzumab).
  Other Names: Tecentriq
Drug: BTCT4465A (Mosunetuzumab) SC — Participants with B-cell NHL and CLL will receive BTCT4465A (Mosunetuzumab) via SC injection.

SUMMARY:
This is a Phase 1/2 dose-escalation study of BTCT4465A (Mosunetuzumab) administered as a single agent and in combination with atezolizumab in participants with relapsed or refractory B-cell NHL and CLL. The study will consist of a dose-escalation stage and an expansion stage where participants will be enrolled into indication-specific cohorts.

ELIGIBILITY:
Key Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* B-cell hematologic malignancies expected to express the cluster of differentiation 20 (CD20) antigen who have relapsed after or failed to respond to at least one prior treatment regimen and for whom there is no available therapy expected to improve survival
* Adequate hepatic, hematologic, and renal function

Key Exclusion Criteria:

* Pregnant or lactating women
* Monoclonal antibody, radioimmunoconjugate, antibody-drug conjugate, chemotherapy, or other investigational anti-cancer agent within 4 weeks prior to study drug
* Treatment with radiotherapy within 2 weeks prior to the first BTCT4465A (Mosunetuzumab) administration
* Systemic immunosuppressive medication within 2 weeks prior to study drug
* Autologous stem cell transplantation (SCT) within 100 days prior to study drug, or any prior allogeneic SCT or solid organ transplantation
* Autoimmune disease with the exception of controlled/treated hypothyroidism, disease-related immune thrombocytopenic purpura, or hemolytic anemia
* History of central nervous system (CNS) lymphoma or other CNS disease
* Significant cardiovascular or pulmonary disease
* Hepatitis B or C or human immunodeficiency virus (HIV)
* Receipt of a live attenuated vaccine within 4 weeks prior to study drug
* Prior treatment with chimeric antigen receptor T-cell (CAR-T) therapy within 30 days before first BTCT4465A (Mosunetuzumab) administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 713 (Actual)
Dates: Start 2015-09-15 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of BTCT4465A (Mosunetuzumab) | BTCT4465A (Mosunetuzumab) single agent: Cycle 1; BTCT4465A (Mosunetuzumab) in combination with atezolizumab: during the first cycle that BTCT4465A (Mosunetuzumab) and atezolizumab are administered concurrently (cycle length = 21 days)
Percentage of Participants With Adverse Events | Cycle 1 Day 1 until 90 days after the last infusion (cycle length = 21 days; up to approximately 14 months)
BTCT4465A (Mosunetuzumab) Serum Concentration | Baseline up to 30 days after the last infusion of BTCT4465A (Mosunetuzumab) (up to approximately 12 months)
Atezolizumab Serum Concentration | Baseline up to 30 days after the last infusion of BTCT4465A (Mosunetuzumab) (up to approximately 12 months)
Percentage of Participants with Complete Response as Assessed Using Standard Criteria for NHL | Baseline up to approximately 4 years (assessed at screening and then every 3 months until disease progression, start of new anti-cancer therapy, or withdrawal)

SECONDARY OUTCOMES:
Duration of Response as Assessed Using Standard Criteria for NHL | Baseline up to approximately 4 years (assessed at screening and then every 3 months until disease progression, start of new anti-cancer therapy, or withdrawal)
Progression-Free Survival (PFS) as Assessed Using Standard Criteria for NHL | Baseline up to approximately 4 years (assessed at screening and then every 3 months until disease progression, start of new anti-cancer therapy, withdrawal, or death from any cause)
Overall Survival | Baseline until death from any cause (up to approximately 4 years)
European Organisation for Research and Treatment of Cancer Quality-of-Life Questionnaire Core 30 (EORTC QLQ-C30) Scores to Assess Health-Related Quality of Life (HRQoL) | Baseline until disease progression, start of new anti-cancer therapy, or withdrawal (up to approximately 4 years).
  The Functional Assessment of Cancer Therapy-Lymphoma (FACT-lym) Subscale, and the EuroQol 5 Dimension-5 Level (EQ-5D-5L) Questionnaire scores will also be used to assess HRQoL
Objective Response Rate (ORR) | Baseline up to approximately 4 years (assessed at screening and then every 3 months until disease progression, start of new anti-cancer therapy, or withdrawal)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (35):
- United States (12):
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - Sansum Medical Clinic, Inc., Santa Barbara, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Yale University School Of Medicine, New Haven, Connecticut
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center - Commack, Commack, New York
  - Memorial Sloan Kettering Cancer Center at Westchester, Harrison, New York
  - New York Uni Medical Center, New York, New York
  - Willamette Valley Cancer Insitute and Research Center, Springfield, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
- Australia (8):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Icon Cancer Care South Brisbane, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - St. Vincent's Hospital Melbourne, Fitzroy, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Monash Health Clinical Trial Pharmacy department, Clayton, Victoria
  - The Perth Blood Institute, Nedlands, Western Australia
- Canada (2):
  - Princess Margaret Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Germany (4):
  - Universitatsklinikum Koln, Cologne
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz
  - Klinikum der Universität München, Campus Großhadern, München
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (4):
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitario Vall d Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Complejo Asistencial Universitario de Salamanca, Salamanca
- United Kingdom (3):
  - Barts Cancer Institute, London
  - The Christie NHS Foundation Trust, Manchester
  - Royal Marsden Hospital;Institute of Cancer Research, Sutton

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing.

REFERENCES:
- [Derived] Lewis KL, Assouline SE, Baker RI, Bartlett NL, El-Sharkawi D, Giri P, Ku M, Matasar MJ, Schuster SJ, Radford J, Wei MC, Yin S, Kwan A, To I, Raghavan V, Budde LE, Cheah CY. Mosunetuzumab monotherapy is active and tolerable in patients with relapsed/refractory Richter's transformation. Blood Adv. 2026 Feb 5:bloodadvances.2025017914. doi: 10.1182/bloodadvances.2025017914. Online ahead of print. PMID 41643182
- [Derived] Danilov AV, Kambhampati Thiruvengadam S, Linton K, Cumings K, Chirikov V, Mutebi A, Bains Chawla S, Chhibber A, Rivas Navarro F, Marques Goncalves F, Wang A, Ding Z, Alshreef A, Favaro E, Hoehn D, Sureda A. Indirect comparison of epcoritamab vs chemoimmunotherapy, mosunetuzumab, or odronextamab in follicular lymphoma. Blood Adv. 2025 Aug 12;9(15):3754-3765. doi: 10.1182/bloodadvances.2024015274. PMID 40472301
- [Derived] Li J, Liao MZ, Wilkins J, Penuel E, Wang B, Vadhavkar S, Peng K, Cao J, Li Z, Zhang Y, Li W, Li D, Zhou M, Wei MC, Kwan A, Zhao R, Li C, Li CC, Turner DC. Ethnic Sensitivity Assessment of Mosunetuzumab Pharmacokinetics and Pharmacodynamics in Chinese Patients With Relapsed or Refractory Follicular Lymphoma. Clin Transl Sci. 2025 May;18(5):e70211. doi: 10.1111/cts.70211. PMID 40279333
- [Derived] Chong EA, Penuel E, Napier EB, Lundberg RK, Budde LE, Shadman M, Matasar MJ, Bartlett NL, Flinn IW, Bosch F, Fay K, Goy A, Kumar A, Nastoupil LJ, Wei MC, Wu M, Yin S, Fraietta JA, Chong ER, Schuster SJ. Impact of prior CAR T-cell therapy on mosunetuzumab efficacy in patients with relapsed or refractory B-cell lymphomas. Blood Adv. 2025 Feb 25;9(4):696-703. doi: 10.1182/bloodadvances.2024013640. PMID 39571171
- [Derived] Sehn LH, Bartlett NL, Matasar MJ, Schuster SJ, Assouline SE, Giri P, Kuruvilla J, Shadman M, Cheah CY, Dietrich S, Fay K, Ku M, Nastoupil LJ, Wei MC, Yin S, To I, Kaufman D, Kwan A, Penuel E, Bolen CR, Budde LE. Long-term 3-year follow-up of mosunetuzumab in relapsed or refractory follicular lymphoma after >/=2 prior therapies. Blood. 2025 Feb 13;145(7):708-719. doi: 10.1182/blood.2024025454. PMID 39447094
- [Derived] Ray MD, Kanters S, Beygi S, Best T, Wulff J, Limbrick-Oldfield E, Patel AR, Oluwole OO. Matching-Adjusted Indirect Comparisons of Axicabtagene Ciloleucel to Mosunetuzumab for the Treatment of Relapsed/Refractory Follicular Lymphoma. Transplant Cell Ther. 2024 Sep;30(9):885.e1-885.e11. doi: 10.1016/j.jtct.2024.06.016. Epub 2024 Jun 19. PMID 38901633
- [Derived] Jemaa S, Ounadjela S, Wang X, El-Galaly TC, Kostakoglu L, Knapp A, Ku G, Musick L, Sahin D, Wei MC, Yin S, Bengtsson T, De Crespigny A, Carano RAD. Automated Lugano Metabolic Response Assessment in 18F-Fluorodeoxyglucose-Avid Non-Hodgkin Lymphoma With Deep Learning on 18F-Fluorodeoxyglucose-Positron Emission Tomography. J Clin Oncol. 2024 Sep 1;42(25):2966-2977. doi: 10.1200/JCO.23.01978. Epub 2024 Jun 6. PMID 38843483
- [Derived] Bender B, Li CC, Marchand M, Turner DC, Li F, Vadhavkar S, Wang B, Deng R, Lu J, Jin J, Li C, Yin S, Wei M, Chanu P. Population pharmacokinetics and CD20 binding dynamics for mosunetuzumab in relapsed/refractory B-cell non-Hodgkin lymphoma. Clin Transl Sci. 2024 Jun;17(6):e13825. doi: 10.1111/cts.13825. PMID 38808543
- [Derived] Budde LE, Assouline S, Sehn LH, Schuster SJ, Yoon SS, Yoon DH, Matasar MJ, Bosch F, Kim WS, Nastoupil LJ, Flinn IW, Shadman M, Diefenbach C, Cheah CY, Ma CY, Huang H, Kwan A, Wei MC, Yin S, Bartlett NL. Durable Responses With Mosunetuzumab in Relapsed/Refractory Indolent and Aggressive B-Cell Non-Hodgkin Lymphomas: Extended Follow-Up of a Phase I/II Study. J Clin Oncol. 2024 Jul 1;42(19):2250-2256. doi: 10.1200/JCO.23.02329. Epub 2024 Mar 28. PMID 38547425
- [Derived] Schuster SJ, Huw LY, Bolen CR, Maximov V, Polson AG, Hatzi K, Lasater EA, Assouline SE, Bartlett NL, Budde LE, Matasar MJ, Koeppen H, Piccione EC, Wilson D, Wei MC, Yin S, Penuel E. Loss of CD20 expression as a mechanism of resistance to mosunetuzumab in relapsed/refractory B-cell lymphomas. Blood. 2024 Feb 29;143(9):822-832. doi: 10.1182/blood.2023022348. PMID 38048694
- [Derived] Bosch F, Kuruvilla J, Vassilakopoulos TP, Maio DD, Wei MC, Zumofen MB, Nastoupil LJ. Indirect Treatment Comparisons of Mosunetuzumab With Third- and Later-Line Treatments for Relapsed/Refractory Follicular Lymphoma. Clin Lymphoma Myeloma Leuk. 2024 Feb;24(2):105-121. doi: 10.1016/j.clml.2023.09.007. Epub 2023 Sep 28. PMID 37981564
- [Derived] Sanchez Alvarez J, Jaber M, Blanchet Zumofen MH. Multiple Real-World Data Sources in a Bayesian Framework to Inform Long-Term Survival Estimates of Mosunetuzumab in Patients with Follicular Lymphoma. Oncol Ther. 2023 Dec;11(4):495-511. doi: 10.1007/s40487-023-00245-4. Epub 2023 Oct 18. PMID 37851321
- [Derived] Bartlett NL, Assouline S, Giri P, Schuster SJ, Cheah CY, Matasar M, Gregory GP, Yoon DH, Shadman M, Fay K, Yoon SS, Panizo C, Flinn I, Johnston A, Bosch F, Sehn LH, Wei MC, Yin S, To I, Li CC, Huang H, Kwan A, Penuel E, Budde LE. Mosunetuzumab monotherapy is active and tolerable in patients with relapsed/refractory diffuse large B-cell lymphoma. Blood Adv. 2023 Sep 12;7(17):4926-4935. doi: 10.1182/bloodadvances.2022009260. PMID 37067952
- [Derived] Budde LE, Sehn LH, Matasar M, Schuster SJ, Assouline S, Giri P, Kuruvilla J, Canales M, Dietrich S, Fay K, Ku M, Nastoupil L, Cheah CY, Wei MC, Yin S, Li CC, Huang H, Kwan A, Penuel E, Bartlett NL. Safety and efficacy of mosunetuzumab, a bispecific antibody, in patients with relapsed or refractory follicular lymphoma: a single-arm, multicentre, phase 2 study. Lancet Oncol. 2022 Aug;23(8):1055-1065. doi: 10.1016/S1470-2045(22)00335-7. Epub 2022 Jul 5. PMID 35803286
- [Derived] Budde LE, Assouline S, Sehn LH, Schuster SJ, Yoon SS, Yoon DH, Matasar MJ, Bosch F, Kim WS, Nastoupil LJ, Flinn IW, Shadman M, Diefenbach C, O'Hear C, Huang H, Kwan A, Li CC, Piccione EC, Wei MC, Yin S, Bartlett NL. Single-Agent Mosunetuzumab Shows Durable Complete Responses in Patients With Relapsed or Refractory B-Cell Lymphomas: Phase I Dose-Escalation Study. J Clin Oncol. 2022 Feb 10;40(5):481-491. doi: 10.1200/JCO.21.00931. Epub 2021 Dec 16. PMID 34914545